CLINICAL TRIAL: NCT02356406
Title: Celiac Plexus Radiosurgery for Pain Management in Advanced Cancer Patients - a Phase II Trial
Brief Title: Celiac Plexus Radiosurgery for Pain Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, David Hausner M.D, palliative care physician, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHEBA-14-1630-DH-CTIL
Record Dates: First submitted 2015-01-21; First posted 2015-02-05 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Digestive System Neoplasms
Keywords: Radiosurgery; Celiac Plexus; Pain; Quality of Life
MeSH Terms: conditions — Digestive System Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celiac Plexus Radiosurgery (Experimental): The study has a prospective, single arm design. It will be composed from an initial run-in safety assessment that will include 6 patients and then continue as a phase II trial.
  All eligible patients will receive the same protocol of celiac plexus radiosurgery
  Interventions: Radiation: Celiac Plexus Radiosurgery

INTERVENTIONS:
Radiation: Celiac Plexus Radiosurgery — 5 fractions of SBRT (Stereotactic body radiation therapy). The target will always include the anterior-medial aspect aorta at T12-L2 (surrogate for celiac plexus). If there is adjacent tumor (e.g. pancreatic tumor that infiltrates the celiac plexus) this will be irradiated in addition.
  It is expected that patients will be treated with a rapid-arc IMRT (Intensity modulation radiation therapy) dose-painting technique. Details of beam arrangement and energy used will be determined on an individual basis.

SUMMARY:
This prospective study evaluates celiac plexus radiosurgery for pain control in patients with upper abdominal malignancies.

DETAILED DESCRIPTION:
This study aims as primary objective to evaluate short and long term pain relief following the administration of radiosurgery to the celiac plexus in patients with upper abdominal cancer. As secondary objectives it will describe acute and late side effects and quality of life measures of patients undergoing the treatment.

The study has a prospective, single arm design. It will be composed from an initial run-in safety assessment that will include 6 patients and then continue as a phase II trial. All eligible patients will receive the same protocol of celiac plexus radiosurgery and will be evaluated before, during and following this treatment.

The treatment duration is one and a half weeks (5 fractions delivered every other weekday).

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper abdominal cancer (pancreatic/gastric/colon/hepato-biliary cancer) with typical retroperitoneal pain syndrome (somatic pain that radiates from the upper abdomen to the back) thought to be secondary to celiac plexus involvement, directly or indirectly, and have high level of pain despite opioids usage (NRS >4). Patients with other cancer types metastatic to the celiac lymph nodes will also be eligible
* Recent abdominal imaging (CT, PET or MRI) should be at most 2 months old.
* Prior chemotherapy or biological treatment is allowed, but any active oncological treatment should be stopped at least 1 week prior to radiation and renewed at least 1 week following radiation. Following gemcitabine 2 weeks are required between final dose and commencement of radiation
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Patients under 18 years of age
* Patients who are well balanced in terms of pain control
* Patients with life expectancy <8 weeks
* Patients with ECOG (Eastern cooperative oncology group) performance status 4
* Any concurrent chemotherapy or biologic treatment is prohibited during 1 week before until 1 week following radiotherapy
* Special populations: pregnant women, prisoners, patients with major psychiatric illnesses
* Previous radiotherapy to upper abdomen
* Conditions associated with increased side effects to radiotherapy (IBD (inflammatory bowel disease) for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain score difference from baseline | 3 weeks post treatment

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) pain score difference from baseline | 6 weeks and 3 months post treatment and subsequently every 3 months on average up to 1 year post treatment
Analgesic use difference from baseline in oral morphin equivalents | 6 weeks and 3 months post treatment and subsequently every 3 months on average up to 1 year post treatment
  Average analgesic consumption will be defined using daily oral morphine equivalents in milligrams
QoL difference from baseline | 6 weeks and 3 months post treatment and subsequently every 3 months on average up to 1 year post treatment
Safety profile of the procedure - measuring the frequency and severity of treatment side effects, mainly GI toxicities | 6 weeks and 3 months post treatment and subsequently every 3 months on average up to 1 year post treatment
  The safety profile will focused on fatigue and expected GI (gastro-intestinal) toxicities as nausea, vomiting and diarrhea. Acute and late toxicity will be assessed using the NCI-CTCAE (common toxicity criteria for adverse events) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: David Hausner, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Levy MJ, Wiersema MJ. EUS-guided celiac plexus neurolysis and celiac plexus block. Gastrointest Endosc. 2003 Jun;57(7):923-30. doi: 10.1016/s0016-5107(03)70036-4. No abstract available. PMID 12776048
- [Background] Kambadakone A, Thabet A, Gervais DA, Mueller PR, Arellano RS. CT-guided celiac plexus neurolysis: a review of anatomy, indications, technique, and tips for successful treatment. Radiographics. 2011 Oct;31(6):1599-621. doi: 10.1148/rg.316115526. PMID 21997984
- [Background] Zhu Z, Friess H, diMola FF, Zimmermann A, Graber HU, Korc M, Buchler MW. Nerve growth factor expression correlates with perineural invasion and pain in human pancreatic cancer. J Clin Oncol. 1999 Aug;17(8):2419-28. doi: 10.1200/JCO.1999.17.8.2419. PMID 10561305
- [Background] Wong GY, Schroeder DR, Carns PE, Wilson JL, Martin DP, Kinney MO, Mantilla CB, Warner DO. Effect of neurolytic celiac plexus block on pain relief, quality of life, and survival in patients with unresectable pancreatic cancer: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1092-9. doi: 10.1001/jama.291.9.1092. PMID 14996778
- [Background] Smigielski J, Piskorz L, Wawrzycki M, Kutwin L, Misiak P, Brocki M. Assessment of quality of life in patients with non-operated pancreatic cancer after videothoracoscopic splanchnicectomy. Wideochir Inne Tech Maloinwazyjne. 2011 Sep;6(3):132-7. doi: 10.5114/wiitm.2011.24690. Epub 2011 Sep 30. PMID 23255971
- [Background] Didolkar MS, Coleman CW, Brenner MJ, Chu KU, Olexa N, Stanwyck E, Yu A, Neerchal N, Rabinowitz S. Image-guided stereotactic radiosurgery for locally advanced pancreatic adenocarcinoma results of first 85 patients. J Gastrointest Surg. 2010 Oct;14(10):1547-59. doi: 10.1007/s11605-010-1323-7. Epub 2010 Sep 14. PMID 20839073
- [Background] Rwigema JC, Parikh SD, Heron DE, Howell M, Zeh H, Moser AJ, Bahary N, Quinn A, Burton SA. Stereotactic body radiotherapy in the treatment of advanced adenocarcinoma of the pancreas. Am J Clin Oncol. 2011 Feb;34(1):63-9. doi: 10.1097/COC.0b013e3181d270b4. PMID 20308870
- [Background] Macchia G, Morganti AG, Cilla S, Ippolito E, Massaccesi M, Picardi V, Mattiucci GC, Bonomo P, Tambaro R, Pacelli F, Piermattei A, De Spirito M, Valentini V, Cellini N, Deodato F. Quality of life and toxicity of stereotactic radiotherapy in pancreatic tumors: a case series. Cancer Invest. 2012 Feb;30(2):149-55. doi: 10.3109/07357907.2011.640649. PMID 22250589
- [Background] Chuong MD, Springett GM, Freilich JM, Park CK, Weber JM, Mellon EA, Hodul PJ, Malafa MP, Meredith KL, Hoffe SE, Shridhar R. Stereotactic body radiation therapy for locally advanced and borderline resectable pancreatic cancer is effective and well tolerated. Int J Radiat Oncol Biol Phys. 2013 Jul 1;86(3):516-22. doi: 10.1016/j.ijrobp.2013.02.022. Epub 2013 Apr 5. PMID 23562768
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Iwata K, Yasuda I, Enya M, Mukai T, Nakashima M, Doi S, Iwashita T, Tomita E, Moriwaki H. Predictive factors for pain relief after endoscopic ultrasound-guided celiac plexus neurolysis. Dig Endosc. 2011 Apr;23(2):140-5. doi: 10.1111/j.1443-1661.2010.01046.x. Epub 2010 Dec 7. PMID 21429019
- [Derived] Hammer L, Hausner D, Ben-Ayun M, Shacham-Shmueli E, Morag O, Margalit O, Boursi B, Yarom N, Jacobson G, Katzman T, Abrams R, Dicker A, Golan T, Symon Z, Lawrence YR. Single-Fraction Celiac Plexus Radiosurgery: A Preliminary Proof-of-Concept Phase 2 Clinical Trial. Int J Radiat Oncol Biol Phys. 2022 Jul 1;113(3):588-593. doi: 10.1016/j.ijrobp.2022.02.038. Epub 2022 Mar 4. PMID 35257800